CLINICAL TRIAL: NCT05702645
Title: Chronic Health Conditions in Down Syndrome-Associated Acute Leukemia: The Down Syndrome Phenotyping Acute Leukemia Study in Survivors (DS-PALS Survivors)
Brief Title: A Study to Learn More About the Health of Persons With Down Syndrome After Treatment for Acute Leukemia
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: ALTE22C1; NCI-2022-09410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE22C1 (Other: Children's Oncology Group); COG-ALTE22C1 (Other: DCP); ALTE22C1 (Other: CTEP); R01CA263000 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: B Acute Lymphoblastic Leukemia Associated With Down Syndrome; Down Syndrome; Myeloid Leukemia Associated With Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Specimen Handling; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood/saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (biospecimen collection, clinical evaluation): Patients undergo an optional saliva/buccal swab in part 1 and clinical assessment in part 2 of the study. Patients with DS-ALL may then undergo blood sample collection and neurocognitive assessment in part 3 of the study.
  Interventions: Procedure: Biospecimen Collection; Other: Clinical Evaluation; Other: Neurocognitive Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Patients undergo saliva/buccal and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Clinical Evaluation — Undergo a clinical assessment
  Other Names: Clinical Assessment
Other: Neurocognitive Assessment — Undergo neurocognitive assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This study attempts to learn more about the health of persons with Down syndrome after treatment for acute leukemia. Children with Down syndrome are at increased risk for side effects during treatment for acute leukemia, but it is unclear of their risk for long-term effects of cancer treatment. By learning more about the factors that may contribute to chronic health conditions and long-term effects after treatment for leukemia in persons with Down syndrome, clinical practice guidelines for survivorship care can be developed to help improve their quality-of-life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the prevalence, type, and severity of chronic health conditions (CHC) in survivors of Down syndrome-associated acute leukemia (DS-AL), and to compare CHC with frequency-matched DS individuals that have no cancer history.

SECONDARY OBJECTIVES:

I. To characterize post-treatment clinical outcomes of DS-AL by prospective, in-person assessment.

II. To determine the prevalence and severity of parent-reported adverse neuropsychological (NP) outcomes in survivors of DS-AL, compared with frequency-matched DS individuals with no cancer history.

III. To determine health-related quality of life (HRQOL) in survivors of DS-AL, compared with frequency-matched DS individuals with no cancer history.

IV. To identify clinical risk determinants of CHC, NP, and clinical outcomes in survivors of DS-AL.

V. To establish a well-annotated cohort of survivors of DS-AL and associated biobank as a resource for future investigations.

EXPLORATORY OBJECTIVES:

I. For DS-acute lymphoblastic leukemia (DS-ALL), test if structural birth defects and genetic associations with etiology extend to CHC.

II. For DS-ALL, test if telomere length determined by polygenic risk score and telomere flow-fluorescence in situ hybridization (FISH) are associated with outcomes from in-person NP assessment.

OUTLINE:

Patients undergo an optional saliva/buccal swab in part 1 and clinical assessment in part 2 of the study. Patients with DS-ALL may then undergo blood sample collection and neurocognitive assessment in part 3 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >= 6 and < 40 years at the time of enrollment
* A diagnosis of Down syndrome is required, and may include any of the three recognized types: trisomy 21 resulting from chromosomal nondisjunction (most common), translocation (the patient has 46 chromosomes, but all or part of an additional copy of chromosome 21 is attached to another chromosome), or mosaicism (trisomy 21 that is present in only a fraction of cells)
* All patients must be DS-AL survivors (acute lymphoblastic leukemia [ALL] or acute myeloid leukemia [AML])

  * Note 1: Myeloid leukemia of Down syndrome (ML-DS) is included in the AML category above. Per the World Health Organization (WHO) definition of ML-DS, this diagnosis encompasses both myelodysplastic syndrome (MDS) and overt AML. Also, note that survivors of relapsed disease are eligible, so long as the patient otherwise meets eligibility criteria, i.e., treatment for relapse was completed at least 36 calendar months prior to enrollment and did not include stem cell transplant
  * Note 2: A diagnosis of transient abnormal myelopoiesis (TAM), also known as transient myeloproliferative disease (TMD), is not alone sufficient for inclusion in this study
* Patients must have been treated for ALL or AML

  * Note: History of COG therapeutic trial participation is not required. As a reminder ML-DS would be included under the AML category here above
* All cancer treatment (oral or intravenous) must have been completed at least 36 calendar months prior to enrollment
* Patients must have a life expectancy of > 1 year
* Patient and parent of subject must be either English or Spanish speaking. At least one parent or guardian must be able to read and write in English or Spanish

  * Note: Parents or guardians are responsible for completing all questionnaires, even in the case of subjects that are >= 18 years old
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with history of hematopoietic stem cell transplant (HSCT) are excluded

  * Note: Patients with previous chimeric antigen receptor T-cell (CAR T-cell) therapy, and other cellular cancer therapies can participate, as long as all other eligibility criteria are satisfied
* Patients with a history of cancers prior to their ALL or AML diagnosis are excluded. Patients that developed a subsequent malignant neoplasm following their ALL or AML diagnosis are also excluded

  * Note: Prior history of transient abnormal myelopoiesis is allowed, but is not sufficient for eligibility
* Patients whose parents or guardians are unable to complete the required forms are excluded

Ages: 6 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: DS-AL survivors from the Children's Oncology Group (COG) Registry and Epidemiology protocols or locally from participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence, type, and severity of chronic health conditions (CHC) | Up to study completion
  Summary statistics will be used to characterize the study populations on CHC outcomes. Quantitative data (number of comorbidities) will be summarized using descriptive statistics and correlational techniques. Will use pooled logistic regression to estimate overall response, 95% confidence interval (CI), and p-values for association of acute leukemia (AL) diagnosis with medical record-verified CHC, agnostic of time to CHC. Will use stratified Cox models to refine associations of AL diagnosis with CHC based on time to CHC incidence. Within each age interval, will estimate the hazard ratio, 95% CI, and p-values to report time-dependent effects of AL diagnosis on CHC.

SECONDARY OUTCOMES:
Post-treatment clinical outcomes | Up to study completion
  Summary statistics will be used to characterize the study population on clinical outcomes, by AL subtype and, for each test, the proportion of normal, abnormal, and missing tests.
Prevalence and severity of parent-proxy neuropsychological (NP) outcomes | Up to study completion
  NP outcomes (measured by both parent proxy and direct assessment) will be reported by both raw and normalized scores, and quantitative data summarized using descriptive statistics and correlational techniques. The mean score for each test will be compared between the cohorts using a student t-test (2-sided significance level of 0.05 and equal variance).
Health-related quality of life (HRQOL) | Up to study completion
  HRQOL will be assessed using the Pediatric Quality of Life Inventory. Parents will be asked to scale 23 items comprising four dimensions (Physical, Emotional, Social, and School functioning) on a 5 point unweighted Likert scale. Will use a t-test (or Wilcoxon rank sum test if appropriate) to compare the mean (or median) HRQOL score.
Clinical risk determinants of CHC, NP, and clinical outcomes | Up to study completion
  Will use Cox regression to estimate the hazard ratio and 95% CI for (1) number, severity, and type of CHC, and (2) NP deficits dichotomized as clinically significant impairment yes/no (=< 1.5 standard deviation outside of the mean for the age-normative sample) according to age at diagnosis, years off therapy, sex, race/ethnicity, diagnosis, and treatment exposures.
Well-annotated cohort of Down syndrome phenotyping acute leukemia study (DS-PALS) survivors and associated biobank | Up to study completion
  The number of patients who agree to be in the Biobanking part of the study and have leftover tumor tissue and some normal blood, bone marrow, or other tissue saved for future research.

OTHER OUTCOMES:
Structural birth defects and genetic associations with etiology extending to CHC for Down syndrome acute lymphoblastic leukemia (DS-ALL) | Up to study completion
  Will determine the association between structural birth defects and the number, organ system category, and severity of CHC in DS-PALS survivors. Will use Cox regression to estimate hazard ratio and 95% CI for number, severity, and type of CHC by number of birth defects. Will explore the role of DS-ALL susceptibility variants identified in our genome-wide assessment on DS-associated CHC in survivors. Will use Cox regression to estimate the association between four DS-ALL susceptibility loci (rs58923657 near IKZF1, rs3731249 in CDKN2A, rs7090445 in ARID5B, and rs3781093 in GATA3) and CHC.
Telomere length (TL) determined by polygenic risk score and telomere flow-fluorescence in situ hybridization (FISH) in association with outcomes from in-person NP assessment for DS-ALL | Up to study completion
  Will determine genetically-estimated TL. Will use a multivariable Cox proportional hazard model to estimate hazard ratio, 95% CI for the association between each of nine variants and risk for NP deficit =<1 standard deviation below the mean, and consider the weighted and unweighted risk score from the number of risk alleles present and previously-published beta estimates. For flow-FISH analyses, TL =< 1st percentile is considered 'very short,' as previously defined. Will determine objective responses for NP deficits =< 1.5 standard deviation below the mean for an age-normative sample in subjects with TL > or =< 1st percentile, adjusted for relevant covariates and treatment factors. Will report 95% CI, p values using a Chi square test (two-tailed p-value of 0.05 statistically significant).

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Gramatges, Principal Investigator — Children's Oncology Group
Locations (68):
- United States (67):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Children's Hospital, London, Ontario, Canada